CLINICAL TRIAL: NCT02009293
Title: Observational Study of the Effect of Pirfenidone on Cough in Patients With Idiopathic Pulmonary Fibrosis
Brief Title: The Effect of Pirfenidone on Cough in Patients With Idiopathic Pulmonary Fibrosis
Acronym: Cough-IPF
Status: Completed | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Collaborators: University of Catania (Other); University of Lyon (Other); King's College Hospital NHS Trust (Other); Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Marlies Wijsenbeek, MD PhD, Erasmus Medical Center
Other Study IDs: NL44729.078.13
Record Dates: First submitted 2013-12-01; First posted 2013-12-11 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: idiopathic pulmonary fibrosis; cough; quality of life
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Cough

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Cough IPF: Male and female with idiopathic pulmonary fibrosis and cough and about to start on Pirfenidone according to regular practice will be asked to wear a cough monitor 24 hours before starting Pirfenidone and twice 24 hours while using Pirfenidone. Patients will also be asked to fill in questionnaires about quality of life and cough.
  Interventions: Other: Cough monitor

INTERVENTIONS:
Other: Cough monitor — questionnaires about cough and quality of life
  Other Names: cough monitoring; Leicester Cough Monitor

SUMMARY:
In this study we evaluate the effect of Pirfenidone on cough and quality of life in patients with idiopathic pulmonary fibrosis (IPF) that are treated with Pirfenidone in daily practice. The hypothesis is that Pirfenidone will decrease cough and increase quality of life.

DETAILED DESCRIPTION:
Rationale: Idiopathic Pulmonary Fibrosis (IPF) is a progressive fibrotic lung disease of unknown cause with a median survival of 3-5 years. No curative treatment exists, though in 2011 Pirfenidone was approved for the treatment of IPF as it appeared to slow down the decline in lung function. In patients with IPF, the most common symptoms are cough and breathlessness. Cough is not only a major distressing and disabling symptom but also an independent predictor of disease progression and death in IPF. Recent preliminary data suggest a possible effect of Pirfenidone on cough.

Objective: In this study we want to objectively measure the effect of Pirfenidone on cough in patients with IPF that are treated with Pirfenidone in daily practice .

Study design: This is a prospective, observational, international multicenter study.

Intervention: Objective 24-hour cough frequency will be recorded using the Leicester Cough Monitor (LCM), a validated ambulatory cough monitoring system, prior to starting with Pirfenidone treatment. The cough recording will be repeated at 4 weeks and at 12 weeks during treatment with Pirfenidone. At the days of cough recording, patients will be asked to fill in questionnaires related to cough and to quality of life. Patient will be treated according to normal clinical practice at their Physician's discretion.

Main study parameters/endpoints: The primary endpoint is change in cough frequency measured by the Leicester cough monitor at week 12 compared to baseline. Secondary endpoints look at the relationships between cough, change in cough, quality of life and clinical parameters.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPF according to American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria (5), definite and probable patients will be eligible
* Written informed consent
* Daily cough related to IPF (exclusion of other causes) present > 8 weeks
* cough score on visual analogue scale of ≥ 40 mm.
* Carbon monoxide transfer capacity corrected for hemoglobin (TLCOc) ≥ 30% and Forced Vital Capacity (FVC) ≥ 50%
* Pirfenidone therapy about to be initiated
* if a history positive for Gastro Esophageal Reflux (GER), using proton pump inhibitor (PPI) > 4 weeks

Exclusion Criteria:

* Opiates, antitussive medication, antihistamines, steroids > equivalent of 10 mg prednisone or N-acetylcysteine (NAC) within two weeks before study
* Change of steroid < 10 mg, inhalation steroids within 2 weeks of the study - History of bronchial hyper responsiveness or asthma or relevant airway obstruction (FEV1/FVC < 0.7)
* within 6 weeks of the start signs of respiratory tract infection, change of sputum production and fever.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with IPF about to start on Pirfenidone according to regular practice in the participating University Hospitals
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in cough frequency measured by cough recorder at week 12 compared to baseline | 12 weeks

SECONDARY OUTCOMES:
Impact of cough on quality of life | 12 weeks
Change in cough frequency measured by cough recorder at 4 weeks compared to baseline | 4 weeks

OTHER OUTCOMES:
Change in Leicester Cough Questionnaire at week 12 compared to baseline | 12 weeks
Change in Visual Analogue Score at week 12 compared to baseline | 12 weeks
Change in cough frequency in relation to FVC | 12 weeks
Clinical characteristics predictive of cough response | 12 weeks
Impact of cough on anxiety and depression | 12 weeks
Change in cough frequency in relation to TLCOc | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: M. S. Wijsenbeek, Dr., Study Chair — Erasmus Medical Centre Rotterdam, The Netherlands; C. Vancheri, Prof., Principal Investigator — University of Catania, Italy; V. Cottin, Prof., Principal Investigator — Louis Pradel hospital, Lyon, France; S Birring, Dr., Principal Investigator — Department of Respiratory Medicine,King's College Hospital.Denmark Hill, London; A Russell, Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust; E Renzoni, Dr., Principal Investigator — Royal Brompton & Harefield NHS Foundation Trust
Locations (3):
- University Lyon 1, Louis Pradel hospital, Lyon. FranceService de pneumologie, hôpital Louis Pradel, Lyon, France
- Regional Centre for Rare Lung Disease University of Catania., Catania, Italy
- Erasmus MC Rotterdam, Dep. of Pulmonology, Rotterdam, Netherlands